CLINICAL TRIAL: NCT03749278
Title: Latina Friends Motivating the Soul (ALMA): A Delayed Intervention Control Trial of Program to Reduce Mental Health Disparities in Latina Immigrant Women
Brief Title: Latina Friends Motivating the Soul (ALMA)
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: This record was a placeholder created before trial was conducted. Trial is now described in NCT03545282.
Sponsor: University of Washington (Other)
Collaborators: National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Principal Investigator, India Ornelas, Associate Professor, School of Public Health, University of Washington
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: STUDY00005476; R01MD012230 (NIH)
Record Dates: First submitted 2018-11-13; First posted 2018-11-21 (Actual); Last update posted 2023-05-10 (Actual); Status verified 2023-05

CONDITIONS: Stress; Depression; Anxiety
Keywords: Mental Health; Minority Health; Latina
MeSH Terms: conditions — Depression; Anxiety Disorders; Psychological Well-Being

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: The investigator and outcomes assessor will not have knowledge of the intervention assigned to individual participants
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ALMA Intervention Group (Experimental): Latina Friends Motivating the Soul (ALMA). This group receives the intervention after baseline assessment.
  Interventions: Behavioral: Latina Friends Motivating the Soul (ALMA)
- ALMA Delayed Intervention Control Group (Active Comparator): Latina Friends Motivating the Soul (ALMA). This group receives the intervention six months after the baseline assessment (after the post-intervention, and 3 month assessments have been completed).
  Interventions: Behavioral: Latina Friends Motivating the Soul (ALMA)

INTERVENTIONS:
Behavioral: Latina Friends Motivating the Soul (ALMA) — In a series of 8 weekly sessions, the program uses a group format to teach and encourage women to use coping strategies to reduce depression and anxiety. Over the course of the eight ALMA sessions, 25 women are (1) engaged in activities to identify coping strategies they are currently using and encouraged to continue to use them; (2) introduced to new coping strategies (e.g. mindfulness techniques, increased social ties and social support); and, (3) provided resources for seeking additional help if needed

SUMMARY:
Latina immigrant women are particularly vulnerable to depression and anxiety due to the social and economic stressors they face, including high levels of poverty, low levels of education, family obligations, exposure to violence, and limited access to community resources. ALMA aims to prevent and reduce depression and anxiety among Latina immigrant women. Women attend 8 weekly sessions in a group format to teach and encourage women to use coping strategies to reduce depression and anxiety. The intervention aims to increase participants' social ties and the social support they receive from other Latina immigrant women. The program also helps decrease the stigma associated with mental health and connects women to mental health services when needed.

DETAILED DESCRIPTION:
The proposed study aims to test the efficacy of the Latina Friends Motivating the Soul (ALMA) intervention in a delayed intervention control trial. ALMA is an 8-week program offered in a group format to teach women new coping strategies and enhance their social ties and social support to prevent and reduce their depression and anxiety. Aim 2 is to determine the efficacy of the ALMA intervention to reduce depressive and anxiety symptoms using a delayed intervention control study design. The investigators will recruit women from community-based organizations serving Latino immigrants to participate in the program, which will be offered in community settings. The investigators will assess process outcomes of recruitment, retention, fidelity, and participant satisfaction through observations and in-depth interviews with participants. The investigators will assess the efficacy of the intervention by comparing changes in women's depressive and anxiety symptoms in the intervention and attention control groups at four time points (baseline, 3-month follow-up, 6-month follow-up, and 9-month follow-up). Aim 3 is to assess the potential impact of the intervention on both individual (stigma, stress, coping strategies) and interpersonal (social support, social ties) factors, and whether the impact of the intervention is mediated by these factors. The research team includes investigators in psychology, medicine, social work and public health, as well as community-based organizations serving Latina immigrants. The study uses rigorous methods to test an innovative program that integrates both culturally relevant and evidenced-based strategies to address significant mental health disparities in a high-risk and underserved population. Findings will help inform future research and practice. Given the growth of the Latino population, identifying interventions that reduce mental health disparities among Mexican immigrant women can have a significant public health impact.

ELIGIBILITY:
Inclusion Criteria:

* To be eligible for study participation, participants must be at least 18 years of age, female, speak Spanish, must self-identify as Latina, and have been born outside of the United States

Exclusion Criteria:

* The investigators will screen for and exclude women who currently have high levels of depressive symptoms (as indicated by a score of 20 or higher on the PHQ-9). If women excluded from the study are not already receiving mental health treatment, the will be referred to mental health providers offering low-cost services in Spanish.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Men will not be included in the study. Participation is limited to this population because the research question addressed is relevant only to Latina women and the mental health concerns of this community.
Enrollment: 0 (Actual)
Dates: Start 2018-09-26 (Actual); Primary Completion 2022-01-01 (Actual); Study Completion 2022-05-31 (Estimated)

PRIMARY OUTCOMES:
Depressive Symptoms | Change measure (baseline, 4 months, 6 months, 9 months)
  Frequency of depressive symptoms as measured by the Patient Health Questionnaire 9 (PHQ-9) in the last two weeks. The PHQ-9 is a multipurpose instrument for screening, diagnosing, monitoring and measuring the severity of depression. Scores range from 0 to 27. In general, a total of 10 or above is suggestive of the presence of depression. Depression Severity: 0-4 none, 5-9 mild, 10-14 moderate, 15-19 moderately severe, 20-27 severe.
Anxiety Symptoms | Change measure (baseline, 4 months, 6 months, 9 months)
  Frequency of anxiety symptoms as measured by the General Anxiety Disorders 7 (GAD_&) in the last two weeks. Generalized Anxiety Disorder 7 (GAD-7) is a self-reported questionnaire for screening and severity measuring of generalized anxiety disorder (GAD). Scores range from 0 to 21. Scores ≥10. Anxiety Severity: 1-4 minimal symptoms, 5-9 mild symptoms, 10-14 moderate symptoms, 15-21 severe symptoms

SECONDARY OUTCOMES:
Stress | Change measure (baseline, 4 months, 6 months, 9 months)
  Frequency of perceived stress in the last month. The Perceived Stress Scale (PSS) is a classic stress assessment instrument. Individual scores on the PSS can range from 0 to 40 with higher scores indicating higher perceived stress. Scores ranging from 0-13 would be considered low stress. Scores ranging from 14-26 would be considered moderate stress. Scores ranging from 27-40 would be considered high perceived stress.

CONTACTS AND LOCATIONS:
Overall Officials: India J Ornelas, PhD, MPH, Principal Investigator — University of Washington
Locations (2):
- United States (2):
  - Casa Latina, Seattle, Washington
  - El Centro de la Raza, Seattle, Washington

REFERENCES:
- [Derived] Miranda MM, Rao D, Price C, Gudino J, Perez G, Maurer S, Nelson AK, Perez-Solorio SA, Ornelas IJ. Amigas Latinas Motivando el Alma: Participant Perspectives on an In-Person and Online Implementation of an Intervention to Promote Mental Health in Latina Immigrant Women. Community Ment Health J. 2024 Jul;60(5):908-918. doi: 10.1007/s10597-024-01244-z. Epub 2024 Mar 2. PMID 38430288
- [Derived] Ornelas IJ, Perez G, Maurer S, Gonzalez S, Childs V, Price C, Nelson AK, Perez Solorio SA, Tran A, Rao D. Amigas Latinas Motivando el Alma: In-Person and Online Delivery of an Intervention to Promote Mental Health Among Latina Immigrant Women. J Integr Complement Med. 2022 Oct;28(10):821-829. doi: 10.1089/jicm.2022.0491. Epub 2022 Jun 20. PMID 35723668